CLINICAL TRIAL: NCT06135298
Title: Augmentation of Pertrochanteric Fracture Proximal Femoral Nail Osteosynthesis Using Calcium Sulphate/Hydroxyapatite Combined With Systemic Bisphosphonate - A Pilot Study of the FARE (Fracture Anchorage and Bone REgeneration) Method
Brief Title: FARE Augmentation of Proximal Femoral Fractures With CaS/HA and Systemic ZA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aksaray University (Other)
Collaborators: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Erdem Aras Sezgin, Associate Professor, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/1702
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Trochanteric Fracture of Femur; Osteoporotic Fracture of Femur; Hip Fractures; Bone Density, Low
Keywords: Proximal femoral nail (PFN); Biphasic apatite sulphate ceramic; Zoledronic acid; Augmentation; Bone regeneration
MeSH Terms: conditions — Hip Fractures; Bone Diseases, Metabolic | interventions — Fracture Fixation, Internal; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: A total of 20 eligible patients with osteoporotic per trochanteric fractures, that are scheduled to be treated with proximal femoral nail (PFN), will be included in the study after informed and approved consent and will be randomized into two groups. Randomization will be performed by the principal investigator, by sealed envelopes, after determining if the patient fulfills the inclusion criteria.
Who Masked: Participant, Investigator
Masking Description: Patients in the study group and the control group will be blind to the group they are assigned to until the end of the trial. As intervention is performed during the surgery, blinding will not be possible for the surgical team. Investigators will be blinded during all evaluations, however due to radio-opaque nature of CERAMENT™ BVF, detection of intervention group is possible in CT, DEXA and X-ray evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OSTEOSYNTHESIS + SYSTEMIC ZOLEDRONIC ACID (Active Comparator): After osteosynthesis, systemic Zoledronic acid 5mg will be given intravenously at day 5 after surgery, during hospitalization.
  Interventions: Procedure: OSTEOSYNTHESIS; Drug: Zoledronic acid
- OSTEOSYNTHESIS + LOCAL CERAMENT BONE VOID FILLER (BVF) + SYSTEMIC ZOLEDRONIC ACID (Experimental): During osteosynthesis, cerament BVF will be used for the augmentation of the helical blade. Then, systemic Zoledronic acid 5mg will be given intravenously at day 5 after surgery, during hospitalization.
  Interventions: Procedure: OSTEOSYNTHESIS; Drug: Zoledronic acid; Device: CERAMENT BONE VOID FILLER (BVF)

INTERVENTIONS:
Procedure: OSTEOSYNTHESIS — Routine procedure for anesthesia and infection prophylaxis according to written instructions will be followed in every patient. The patient will be operated supine with the fractured leg positioned in traction table. The hip region is scrubbed and dressed in sterile drapes. Using standard technique, a nail is inserted into the intramedullary canal after fracture reduction. To insert the helical blade in the femoral neck, 2.0 mm diameter guide wire is first placed in the femoral neck, checking the fluoroscopic AP and lateral views. The canal is opened using a 10 mm drill bit and the length of helical blade is measured. After the pilot hole is created for the helical blade placement, the hollow helical blade will be inserted to its end position with gentle blows with a hammer.
  Other Names: Proximal femoral nail with helical blade
Drug: Zoledronic acid — Zoledronic acid (ZA), is a bisphosphonate, and has been shown to reduce the risk of hip fracture by 41% in post-menopausal women. For systemic injection, 5 mg (as per clinical protocol) will be injected intravenously 5 days after surgery, during hospitalization.
  Other Names: Ronidro 5mg/Bag 100 mL Inj
Device: CERAMENT BONE VOID FILLER (BVF) — In addition to the standard surgical procedure, in the study group, after creating the canal with 10 mm drill bit and partly insertion of the helical blade, the synthetic bone void filler CaS/HA will be injected. The helical blade will be inserted partially with gentle blows with a hammer, 2.5 cm from its final intended position. The injectable CaS/HA biomaterial will be mixed as per the manufacturer guidelines and the paste will be transferred into an injection syringe. At t = 2.5 min from the start of mixing, 2-3 mL of BVF paste will be injected by a CE marked Introducer Needle connected to the injection syringe, through the hollow helical blade. Finally, the helical blade will be inserted to its end position with gentle blows with a hammer. Remaining material approximately 2 mL still being moldable will be manually deposited in the trochanteric fracture void.
  Other Names: CaS/HA
  Arms: OSTEOSYNTHESIS + LOCAL CERAMENT BONE VOID FILLER (BVF) + SYSTEMIC ZOLEDRONIC ACID

SUMMARY:
The goal of this clinical trial is to investigate the new bone formation around a metal device in the femoral head in patients with osteoporotic hip fractures undergoing surgical treatment with nails. These surgeries have a high risk of fixation failure in patients with osteoporosis due to low bone quality. The main question we aim to answer are whether promoting new bone formation around the implant is possible with a bone graft substitute (CERAMENT™ Bone Void Filler) and systemic osteoporosis drug (zoledronic acid) combination, which can strengthen the surgical fixation of the fracture. Participants will consist of patients suffering hip fracture and already scheduled for surgical treatment with a nail. One group will undergo conventional surgery. While the other group will also undergo the same surgery, they will receive CERAMENT™ Bone Void Filler around the implant as a short, extra step during surgery. This will allow the researchers to see whether new bone is formed during a 6-month follow-up.

DETAILED DESCRIPTION:
A total of 20 eligible patients with osteoporotic per trochanteric fractures, that are treated with proximal femoral nail (PFN), will be included in the study after informed and approved consent and will be randomized into two groups. Randomization will be performed by the principal investigator, by sealed envelopes, after determining if the patient fulfills the inclusion criteria.

Following randomization, all patients will be operated with PFN. The control group will receive a standard surgical procedure without augmentation of the helical blade. The study group will also receive 2-3 mL of CERAMENT™ BONE VOID FILLER (510(k) Number K201535) delivered using an introducer needle inserted through the helical blade of the PFN inserted in the femoral head, away from the fracture site, with an intent to increase bone-implant anchorage.

Routine procedure for anesthesia and infection prophylaxis according to written instructions will be followed in every patient. For infection infection prophylaxis, 2g cefazolin will be administered 1 hour preoperatively as well as 100 mg doyxcycline 2 hours preoperatively and 6 hours postoperatively. The patient will be operated supine with the fractured leg positioned in traction table. In the standard protocol, fluoroscopy is used to get AP and lateral view during surgery. The hip region is scrubbed and dressed in sterile drapes. Using standard technique, a nail is inserted into the intramedullary canal after fracture reduction. To insert the helical blade in the femoral neck, 2.0 mm diameter guide wire is first placed in the femoral neck, checking the fluoroscopic AP and lateral views. The canal is opened using a 10 mm drill bit and the length of helical blade is measured.

In addition to the standard surgical procedure, in the study group, after creating the canal with 10 mm drill bit and partly insertion of the helical blade, the synthetic bone void filler Calcium Sulphate/Hydroxyapatite (CaS/HA) will be injected.

After the pilot hole is created for the helical blade placement, the hollow helical blade will be inserted partially with gentle blows with a hammer, 2.5 cm from its final intended position. At this point, the injectable CaS/HA biomaterial will be mixed as per the manufacturer guidelines and the paste will be transferred into an injection syringe. At t = 2.5 min from the start of mixing, 2-3 mL of bone void filler (BVF) paste will be injected by a CE marked Introducer Needle connected to the injection syringe, through the hollow helical blade. Under fluoroscopic guidance, injection will start proximal and continue while the cannula is slowly retracted towards the tip of the helical blade until the drilled space in front of the lag screw and the surrounding cancellous bone is filled with 2-3 mL of the material. Finally, the helical blade will be inserted to its end position with gentle blows with a hammer. Remaining material approximately 2 mL still being moldable will be manually deposited in the trochanteric fracture void. A very similar injection technique for application in a dynamic hip screw (DHS) in trochanteric fractures is described in a recently published scientific article.

Patients with an osteoporotic trochanteric femoral fracture that have no contraindications should receive secondary fracture prevention with a bisphosphonate. In this study, all patients will receive systemic (Intravenous) Zoledronic acid (ZA) as routine. All patients included in the study without any contraindication for ZA, therefore will receive 5mg/100ml ZA intravenously day 5 after surgery, during hospitalization. ZA has been shown to significantly reduce the risk of hip fracture in post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Being between 65-90 years of age at the time of fracture
* Acute, unilateral proximal hip fracture (AO Foundation/Orthopaedic Trauma Association [AO/OTA]: A1 and A2) caused by low energy trauma
* Physical condition eligible for surgery with proximal femoral nail
* Having low mortality and high fracture risk according to Fracture and Mortality Risk Evaluation Index (FAME) classification
* Patient with communicative ability to understand the procedure and participate in the study and the follow-up program, consented to be included in the study and signed the consent form

Exclusion Criteria:

* Previous hip or pelvis fracture on the same side
* Concurrent corticosteroid treatment
* Concurrent medical osteoporosis treatment
* Irreversible coagulopathy or bleeding disorder.

  o Note regarding reversible coagulopathies: Patients on coumadin or other anticoagulants may participate. Investigators will follow routine practices for perioperative discontinuation and re-initiation of anti-coagulants.
* Concurrent dialysis or elevated creatinine
* Presence of hypo- or hyper calcaemia
* History or active treatment due to malignancy involving the pelvis/hip area, including ongoing or completed radiotherapy
* Fractures involving acetabulum
* Active systemic infection or local skin infection at the incision site
* Known hyperthyroidism or thyroid adenoma,
* History of serious reaction to iodine-based radio contrast agents
* Patient without communicative ability to understand the procedure and participate in the study and the follow-up program, did not consent to be included in the study and/or did not sign the consent form

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Change of bone density around the helical blade of proximal femoral nail | 1-week and 6 months after the surgery
  Change of bone density measured by Dual-energy X-ray absorptiometry (DEXA) scan of bilateral proximal femurs will be evaluated. A 10 % increase in bone density / bone volume in the femoral head adjacent to the helical blade is expected to be significant and clinically relevant.
Bone remodeling around the helical blade of proximal femoral nail | 1-week and 6 months after the surgery
  Bone remodeling around the helical blade will be evaluated by computerized tomography (CT) scan of the pelvis using a program for alleviating metal artefacts. A 10 % increase in bone density / bone volume in the femoral head adjacent to the helical blade is expected to be significant and clinically relevant.

SECONDARY OUTCOMES:
Harris Hip Score | 1-week and 6 months after the surgery
  The Harris Hip Score (HHS) has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points). The higher the HHS, the less dysfunction. A total score of <70 is considered a poor result; 70-80 is considered fair, 80-90 is good, and 90-100 is an excellent result.
Screw position and migration by X-ray | 1-week and 6 months after the surgery
  X-ray evaluation will quantify helical blade migration on anteroposterior (AP) radiographs by two investigators independently, accounting for femoral rotation and flexion.
Evaluation of fracture union | 6 months after the surgery
  Radiographic evaluation will be performed by two investigators independently to decide whether fracture fixation resulted with union or non-union.
Any mechanical complications | 6 months after the surgery
  Any mechanical complications related to the implant will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Erdem Aras Sezgin, MD, Principal Investigator — Aksaray University
Locations (1):
- Aksaray University Training and Research Hospital, Aksaray, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black DM, Delmas PD, Eastell R, Reid IR, Boonen S, Cauley JA, Cosman F, Lakatos P, Leung PC, Man Z, Mautalen C, Mesenbrink P, Hu H, Caminis J, Tong K, Rosario-Jansen T, Krasnow J, Hue TF, Sellmeyer D, Eriksen EF, Cummings SR; HORIZON Pivotal Fracture Trial. Once-yearly zoledronic acid for treatment of postmenopausal osteoporosis. N Engl J Med. 2007 May 3;356(18):1809-22. doi: 10.1056/NEJMoa067312. PMID 17476007
- [Result] Raina DB, Markeviciute V, Stravinskas M, Kok J, Jacobson I, Liu Y, Sezgin EA, Isaksson H, Zwingenberger S, Tagil M, Tarasevicius S, Lidgren L. A New Augmentation Method for Improved Screw Fixation in Fragile Bone. Front Bioeng Biotechnol. 2022 Mar 2;10:816250. doi: 10.3389/fbioe.2022.816250. eCollection 2022. PMID 35309986
- [Result] Sezgin EA, Tor AT, Markeviciute V, Sirka A, Tarasevicius S, Raina DB, Liu Y, Isaksson H, Tagil M, Lidgren L. A combined fracture and mortality risk index useful for treatment stratification in hip fragility fractures. Jt Dis Relat Surg. 2021;32(3):583-589. doi: 10.52312/jdrs.2021.382. Epub 2021 Nov 19. PMID 34842088